CLINICAL TRIAL: NCT00791804
Title: A Phase II Study Evaluating Inhaled AeroLEF(Liposome-Encapsulated Fentanyl 500mcg/mL)for Post-Operative Pain in Adults After ACL Knee Surgery.
Brief Title: Phase II Study of Inhaled AeroLEF for Analgesia After ACL Knee Surgery
Acronym: Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: YM BioSciences (Industry)
Responsible Party: YM BioSciences Inc.., YM BioSciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLXLEF0
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2008-11-17 (Estimated); Status verified 2008-11

CONDITIONS: Pain; Post Operative Pain
Keywords: Pain; Post Op pain; Fentanyl; Pain Control; Surgery
MeSH Terms: conditions — Pain; Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: AeroLEF

INTERVENTIONS:
Drug: AeroLEF — Inhaled AeroLEF (Liposome-Encapsulated Fentanyl 500 mcg/mL)
  * for nebulized administration as required by the patient.
  * Up to a 6 mL volume (2 x 3 mL doses) containing 500 mcg/ml fentanyl.
  Other Names: Liposome-Encapsulated Fentanyl

SUMMARY:
To evaluate the safety and efficacy of self-titration to effective analgesia with inhaled AeroLEF in patients with moderate/severe acute pain in the post-surgical setting.

DETAILED DESCRIPTION:
After elective ACL knee surgery, consented patients will receive a single dose of AeroLEF for moderate/severe acute pain. Patients stop dosing if they achieve analgesia, complete the maximum available dose, or experience dose-limiting side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between ages 18 years and 60 years.
2. A body mass index of between 18 and 30, inclusive.
3. If a female of child-bearing potential, the patient must have a negative urine pregnancy test at screening and baseline.
4. Scheduled for elective ACL arthroscopic knee repair surgery, and meet the criteria of the American Society of Anesthesiologists [ASA] Physical Status Criteria of Class I or Class II, and suitability for an anesthetic plan limited to general anesthesia (inhalation/IV) with post-operative PCA initiated in a PACU setting and not requiring CPM before the 12 hours post surgery observation is completed.
5. Scheduled for a morning surgery and anticipating remaining in the hospital for an overnight stay.
6. Normal laboratory values for clinical chemistry, haematology and urinalysis. If a patient has abnormal clinically significant laboratory values, inclusion will be permitted at the discretion of the investigator .
7. Physical examination with no clinically relevant findings as determined by the investigator.
8. Able to demonstrate the ability to understand the requirements of the study, willingness to provide written informed consent (prior to any study-related procedures being performed) and able to adhere to the study restrictions, and return for the required assessments.

Exclusion Criteria:

1. History of addiction to drugs or alcohol.
2. Exposure to any investigational drug within the 30 days prior to enrolment.
3. Documented hypersensitivity to fentanyl or other opioid analgesics
4. Documented hypersensitivity/allergy to the components of the liposomes used in the AeroLEF formulation
5. History of pulmonary, cardiovascular, neurologic, endocrine, hepatic, GI, or kidney disease or therapy that would jeopardize the patient's well-being by participation in this study (excluded by ASA I and II categories)
6. Currently receiving treatment, or have received treatment in the previous two weeks, with antidepressant or antipsychotic drugs (including monoamine oxidase inhibitors).
7. Clinically significant ongoing medical conditions.
8. Currently receiving treatment for chronic pain.
9. Current therapy with narcotic or CNS-depressant medications.
10. Current chronic therapy with NSAIDs, ASA or acetaminophen within the previous 7 days.
11. Patient, who in the opinion of the investigator, is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.
12. Blood donation or other blood loss within 45 days prior to enrolment in the study totalling 100 mL or greater.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2004-02; Primary Completion 2004-06 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the time to effective analgesia following initiation of dosing with AeroLEF | Post operative period 12 hours

SECONDARY OUTCOMES:
Time to first perceptible analgesic effect | Post-operative period 12 hours
Time and total of first rescue analgesic | Post-operative period 12 hours
Duration of effective analgesia | Post-operative period 12 hours
Pain rating scores | Post-operative period 12 hours
Adverse events | Post-operative period 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD FRCPC, Principal Investigator — University Health Network, Toronto; Alexander John M Clark, MD FRCPC, Principal Investigator — Queen Elizabeth II Health Sciences Centre
Locations (2):
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre, Capital Health, Halifax, Nova Scotia
  - University Health Network, Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- See also: American Society of Anesthesiologists 2004 Annual Meeting, Abstract A-77 — http://www.asaabstracts.com/strands/asaabstracts/searchresults.htm;jsessionid=3454C2BB815F1946F5043914A5077AE5?base=1&index=1&display=10&highlight=true&highlightcolor=0&bold=true&italic=false